CLINICAL TRIAL: NCT07119060
Title: Monocentric, Controlled, Randomized Trial: Comparison of Pregnancy Rates in Women With One or More Endometriomas, Treated by Cystectomy, Plasma Vaporization, or Sclerotherapy
Brief Title: Ablative Technique For Ovarian Preservation In Endometrioma
Acronym: ATOPE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Tivoli Ducos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CliTiv-01-2025; 2024-A01400-47 (Other: ANSM)
Record Dates: First submitted 2025-07-23; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Endometrioma; Fertility
Keywords: surgery; endometrioma; endometriosis; kystectomy; sclerotherapy; plasma vaporization; fertility
MeSH Terms: conditions — Endometriosis | interventions — Cystectomy; Sclerotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- cystectomy (Experimental): Surgical removal of the endometrioma by gently pulling the cyst wall away from the ovarian tissue (divergent traction technique)
  Interventions: Procedure: Cystectomy
- vaporization with plasma (Active Comparator): It consists of destroying the cyst wall (vaporization) using plasma energy.
  Interventions: Procedure: plasma vaporization
- sclerotherapy (Other): Ethanol sclerotherapy destroys the endometriotic tissue lining the inner wall of the cyst through prolonged contact with 96% ethanol.
  Interventions: Procedure: Sclerotherapy

INTERVENTIONS:
Procedure: Cystectomy — Surgical removal of the endometrioma by gently pulling the cyst wall away from the ovarian tissue (divergent traction technique)
  Arms: cystectomy
Procedure: plasma vaporization — It consists of destroying the cyst wall (vaporization) using plasma energy
  Arms: vaporization with plasma
Procedure: Sclerotherapy — Ethanol sclerotherapy destroys the endometriotic tissue lining the inner wall of the cyst through prolonged contact with 96% alcohol
  Arms: sclerotherapy

SUMMARY:
The goal of this clinical trial is to compare pregnancy rates after different surgical treatments for endometriomas in adult women who have one or more ovarian cysts (endometriomas) larger than 2 cm requiring surgery. The main questions it aims to answer are:

How many women become pregnant within 24 months after surgery ? What are the birth rates and different types of pregnancies (natural, with fertility treatments, and those continuing beyond 12 weeks)? How often do the endometriomas come back after surgery? What surgery-related complications occur? How do pain levels change after treatment?

Researchers will compare different surgical treatment groups to see if one approach results in better pregnancy outcomes and fewer complications.

Participants will:

Be randomly assigned to different surgical treatment groups Undergo surgery for their endometriomas and endometriosis Attend follow-up visits at 3 months and 24 months after the procedure Have their pregnancy outcomes, pain levels, and potential complications monitored throughout the study period

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 18 and 43 years (inclusive)
* Patient diagnosed with endometriosis (by histology or imaging) and symptomatic, requiring surgery (pelvic pain and/or infertility and/or risk to an organ)
* Pelvic MRI or ultrasound performed within the last year showing at least one endometrioma larger than 20 mm in diameter
* Patient with an intention to conceive (probable or certain) after surgery
* Patient informed and having signed the consent form
* Patient covered by a social security scheme

Exclusion Criteria:

* Intraoperative finding that the cyst is not an endometrioma
* Patient under guardianship, conservatorship, or incapable of giving consent
* Patient without sufficient understanding of the French language
* Patient under judicial protection measures
* Patient who is pregnant or breastfeeding

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 332 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2034-07 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
To compare pregnancy rates observed up to 24 months after surgery for endometriosis with endometrioma treatment | From enrollment to 24 months after the surgery
  A Pregnancy is considered if the CGH is >1000 UI/L or a intra uterine pregnancy after 5 weeks of amenorrhea

SECONDARY OUTCOMES:
To compare birth rates pregnancies | From enrollment to 24 months after the surgery
To compare spontaneous pregnancy rates | From enrollment to 24 months after the surgery
To compare pregnancies achieved through assisted reproductive technology (ART) | From enrollment to 24 months after the surgery
To compare pregnancies progressing beyond 12 weeks of amenorrhea | From enrollment to 24 months after the surgery
To compare the recurrence rate of endometriomas, defined as the appearance of an endometrioma larger than 2 cm on the same ovary. | From enrollment to 24 months after the surgery
To compare postoperative complication rates | During 3 months after the surgery
To compare pain scores using the Biberoglu and Behrman scale (Biberoglu and Behrman >4) | From enrollment to 24 months after the surgery
  Pelvic pain will be assessed using the Biberoglu and Behrman scale, which evaluates pain in three domains: dysmenorrhea, dyspareunia, and pelvic pain on palpation. Each domain is scored from 0 (no pain) to 3 (severe pain), with a total score ranging from 0 to 9.
  Higher scores indicate more severe pain (i.e., a worse outcome). A score greater than 4 is considered clinically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Horace ROMAN, Study Director — IFEMEndo - Clinique Tivoli; Adrien CRESTANI, Principal Investigator — IFEMEndo - Clinique Tivoli
Locations (1):
- IFEMEndo - Clinique Tivoli, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie the results reported in this study (after de-identification) will be shared.
Time Frame: The data will be available beginning 12 months after publication of the primary results, for a period of 3 years.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal and whose aims are compatible with the original study objectives